CLINICAL TRIAL: NCT06921473
Title: Effect of Ephedrine and Norepinephrine on Fetal Acidosis During Cesarean Section Under Spinal Anesthesia: A Prospective, Randomized Controlled Trial
Brief Title: Effect of Ephedrine vs. Norepinephrine on Prevention of Fetal Acidosis During Cesarean Section Under Spinal Anesthesia
Acronym: NEO-FET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: mehmet özkılıç (Other)
Responsible Party: Sponsor-Investigator, mehmet özkılıç, Specialist Doctor in Anesthesiology and Reanimation, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Organization: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GYEAH-OB-NE-EF-001
Record Dates: First submitted 2025-04-01; First posted 2025-04-10 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cesarean Delivery Affecting Newborn; Acidosis; Maternal Hypotension; Spinal Aneshtesia
Keywords: Fetal Acidosis; Maternal Hypotension; Ephedrine; Norepinephrine
MeSH Terms: conditions — Acidosis | interventions — Norepinephrine; Ephedrine

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double-blind, two-arm parallel assignment study. Participants are allocated in a 1:1 ratio to receive either ephedrine or norepinephrine intravenously for the prevention of spinal anesthesia-induced hypotension during cesarean section. Randomization is stratified, and the study drugs are prepared and administered in a blinded manner.
Who Masked: Participant
Masking Description: No other parties are masked in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ephedrine Group (Active Comparator): Participants in this group will receive intravenous bolus doses of ephedrine (5-10 mg) to manage spinal anesthesia-induced hypotension during cesarean section.
  Interventions: Drug: Ephedrine
- Norepinephrine Group (Experimental): Participants in this group will receive intravenous bolus doses of norepinephrine (5-10 µg) to manage spinal anesthesia-induced hypotension during cesarean section.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Norepinephrine — Intravenous bolus of norepinephrine (5-10 µg) to treat spinal anesthesia-induced hypotension during cesarean section.
  Other Names: Steradin®
  Arms: Norepinephrine Group
Drug: Ephedrine — Intravenous bolus of 5-10 mg ephedrine administered as needed to treat maternal hypotension following spinal anesthesia during elective cesarean section. The drug is prepared in identical, unlabeled syringes to ensure blinding.
  Other Names: Ephedrine hydrochloride
  Arms: Ephedrine Group

SUMMARY:
This study compares the effects of two medications, ephedrine and norepinephrine, on the baby (fetus) when used to treat low blood pressure (hypotension) during cesarean section under spinal anesthesia. Hypotension is a common side effect during spinal anesthesia, and it can affect the blood flow to the baby. Both medications are commonly used to manage this condition. The goal of the study is to determine which medication is more effective and safer for the baby, by measuring the pH level in the umbilical artery after birth. The study will also examine maternal blood pressure, heart rate, and the baby's Apgar scores.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, controlled clinical trial designed to compare the effects of ephedrine and norepinephrine on fetal acidosis during cesarean section performed under spinal anesthesia. Maternal hypotension is a frequent complication associated with spinal anesthesia, and the management of this condition is critical for maintaining adequate uteroplacental perfusion. While both ephedrine and norepinephrine are commonly used vasopressors, there is ongoing debate regarding their relative safety and efficacy, particularly in terms of fetal outcomes.

The primary aim of this study is to evaluate the incidence of fetal acidosis, defined as an umbilical artery pH < 7.20, in patients receiving either ephedrine or norepinephrine. Secondary outcomes include maternal blood pressure control, heart rate, incidence of maternal and fetal tachycardia, Apgar scores at 1 and 5 minutes, and the need for additional vasopressor support. A total of 100 pregnant women undergoing elective cesarean section will be enrolled, with 50 participants in each treatment group. All participants will receive standardized spinal anesthesia, and vasopressors will be titrated according to protocol.

The study is designed to inform clinical decision-making regarding optimal vasopressor selection in obstetric anesthesia, with a focus on balancing maternal hemodynamic stability and fetal well-being.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged between 18 and 45 years
* Singleton pregnancy at ≥ 37 weeks of gestation
* Scheduled for elective cesarean section under spinal anesthesia
* ASA (American Society of Anesthesiologists) physical status classification I or II
* Ability to understand and sign the informed consent form

Exclusion Criteria:

* History of allergy or hypersensitivity to ephedrine or norepinephrine
* Multiple gestation pregnancies
* Diagnosis of pre-eclampsia, eclampsia, or other hypertensive disorders of pregnancy
* Known cardiovascular disease or arrhythmia
* Placental abnormalities (e.g., placenta previa, placental abruption)
* Fetal structural or chromosomal anomalies
* Morbid obesity (BMI > 40 kg/m²)
* Refusal to participate or inability to provide informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence of fetal acidosis (umbilical artery pH < 7.20) | Within 5 minutes after birth
  Fetal acidosis is defined as an umbilical artery blood pH < 7.20. Arterial blood will be collected from a double-clamped segment of the umbilical cord immediately after delivery and analyzed using a validated blood gas analyzer.

SECONDARY OUTCOMES:
Incidence of maternal hypotension | Within 30 minutes post-spinal anesthesia
  Defined as a decrease in systolic blood pressure >20% from baseline or <90 mmHg. Non-invasive blood pressure is monitored continuously.
Incidence of maternal tachycardia | During surgery
  Maternal tachycardia is defined as a heart rate greater than 100 bpm recorded after vasopressor administration. Heart rate is continuously monitored using ECG. The outcome is the proportion of participants with tachycardia.

OTHER OUTCOMES:
Apgar score at 1 minute | At 1 minute after delivery
  Apgar Score (Appearance, Pulse, Grimace, Activity, Respiration) will be assessed by the attending neonatologist. The score ranges from 0 to 10, where higher scores indicate better neonatal condition. The outcome is the distribution of Apgar scores at 1 minute after birth.
Apgar score at 5 minutes | At 5 minutes after delivery
  Apgar Score (Appearance, Pulse, Grimace, Activity, Respiration) will be assessed by the attending neonatologist. The score ranges from 0 to 10, where higher scores indicate better neonatal condition. The outcome is the distribution of Apgar scores at 5 minutes after birth.
Requirement for additional vasopressor doses | During surgery
  The number and total dosage of additional vasopressor boluses (ephedrine in mg or norepinephrine in µg) required after the initial dose will be recorded for each participant.
Incidence of fetal tachycardia | At delivery
  Fetal tachycardia is defined as a fetal heart rate greater than 160 bpm, assessed using cardiotocography prior to delivery. The outcome is the proportion of fetuses with tachycardia

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet ÖZKILIÇ, Anesthesiology and Intensive Care Specialist, MD, Principal Investigator — Gazi Yaşargil Training and Research Hospital
Locations (1):
- SBÜ Gazi Yaşargil Eğitim ve Araştırma Hastanesi, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because data sharing was not included in the approved study protocol.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-06-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT06921473/Prot_SAP_000.pdf